CLINICAL TRIAL: NCT00091247
Title: An Exploratory, Placebo-Controlled Trial of Prophylactic Tetracycline for Gefitinib-or Cetuximab-Induced Skin Rash (or Other Epidermal Growth Factor Receptor (EGFR) Inhibitor-Induced Skin Rash)
Brief Title: Tetracycline in Preventing Skin Rash in Patients Who Are Receiving Drugs Such as Gefitinib and Cetuximab for Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: NCCTG-N03CB; NCI-2011-01620 (Registry Identifier: CTRP (Clinical Trials Reporting System)); CDR0000385682 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2004-09-07; First posted 2004-09-09 (Estimated); Last update posted 2017-03-16 (Actual); Status verified 2017-03

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — Tetracycline

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- tetracycline (Experimental): Patients receive oral tetracycline twice daily. Treatment continues for 4 weeks in the absence of unacceptable toxicity.
  Quality of life is assessed at baseline and then weekly for 8 weeks.
  Patients are followed at weeks 4 and 8.
  Interventions: Drug: tetracycline hydrochloride
- placebo (Placebo Comparator): Patients receive oral placebo twice daily. Treatment continues for 4 weeks in the absence of unacceptable toxicity.
  Quality of life is assessed at baseline and then weekly for 8 weeks.
  Patients are followed at weeks 4 and 8.
  Interventions: Other: placebo

INTERVENTIONS:
Drug: tetracycline hydrochloride
  Arms: tetracycline
Other: placebo
  Arms: placebo

SUMMARY:
RATIONALE: Tetracycline may be effective in preventing skin rash that is caused by treatment with drugs such as gefitinib or cetuximab.

PURPOSE: This randomized clinical trial is studying tetracycline to see how well it works compared to placebo in preventing skin rash in patients who are receiving drugs such as gefitinib or cetuximab for cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the 1-month incidence and severity of gefitinib-, cetuximab-, or other epidermal growth factor receptor inhibitor-induced skin rash development in patients with cancer treated with tetracycline vs placebo.
* Compare the toxicity of these drugs in these patients.
* Compare the quality of life of patients treated with these drugs who develop vs those who do not develop a rash.
* Determine whether patients who discontinue tetracycline at 1 month develop a rash.

OUTLINE: This is a randomized, double-blind, placebo-controlled, multicenter study. Patients are stratified according to prior chemotherapy regimen (first-line therapy vs other), concurrent epidermal growth factor receptor inhibitor therapy (gefitinib vs cetuximab vs other), and concurrent corticosteroid therapy (yes vs no). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive oral tetracycline twice daily.
* Arm II: Patients receive oral placebo twice daily. In both arms, treatment continues for 4 weeks in the absence of unacceptable toxicity.

Quality of life is assessed at baseline and then weekly for 8 weeks.

Patients are followed at weeks 4 and 8.

PROJECTED ACCRUAL: A total of 126 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of cancer
* Began therapy within the past 7 days or plans to begin therapy within 7 days after study entry with one of the following epidermal growth factor receptor inhibitors:

  * Gefitinib
  * Cetuximab
  * Erlotinib
  * Monoclonal antibody ABX-EGF
  * ICR-62
  * CI-1033
  * EMD-72000
* No rash at study entry

PATIENT CHARACTERISTICS:

Age

* 18 and over

Hepatic

* Bilirubin ≤ 2 mg/dL

Renal

* Creatinine ≤ 2 mg/dL

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective non-hormonal contraception
* Able to take oral medication
* No history of skin condition that may flare during study treatment
* No prior allergic reaction or severe intolerance to tetracycline or one of its derivatives
* No severe nausea or vomiting that would preclude retaining study drug

PRIOR CONCURRENT THERAPY:

Other

* More than 1 week since prior tetracycline
* No milk products, antacids, or calcium supplements for 2 hours before until 2 hours after drug administration
* No other concurrent tetracycline

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2004-12; Primary Completion 2005-08 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Rash severity | Up to 8 weeks
1-month incidence and severity | Up to 8 weeks

SECONDARY OUTCOMES:
quality of life | Up to 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Aminah Jatoi, MD, Study Chair — Mayo Clinic
Locations (69):
- United States (69):
  - Rush-Copley Cancer Care Center, Aurora, Illinois
  - Joliet Oncology-Hematology Associates, Limited - West, Joliet, Illinois
  - Carle Cancer Center at Carle Foundation Hospital, Urbana, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - Saint Anthony Memorial Health Centers, Michigan City, Indiana
  - Cedar Rapids Oncology Associates, Cedar Rapids, Iowa
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Cancer Center of Kansas, PA - Chanute, Chanute, Kansas
  - Cancer Center of Kansas, PA - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, PA - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas, PA - Kingman, Kingman, Kansas
  - Southwest Medical Center, Liberal, Kansas
  - Cancer Center of Kansas, PA - Newton, Newton, Kansas
  - Cancer Center of Kansas, PA - Parsons, Parsons, Kansas
  - Cancer Center of Kansas, PA - Pratt, Pratt, Kansas
  - Cancer Center of Kansas, PA - Salina, Salina, Kansas
  - Cancer Center of Kansas, PA - Wellington, Wellington, Kansas
  - Associates in Womens Health, PA - North Review, Wichita, Kansas
  - Cancer Center of Kansas, PA - Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas, PA - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Cancer Center of Kansas, PA - Winfield, Winfield, Kansas
  - Hickman Cancer Center at Bixby Medical Center, Adrian, Michigan
  - Saint Joseph Mercy Cancer Center, Ann Arbor, Michigan
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - Oakwood Cancer Center at Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - Foote Memorial Hospital, Jackson, Michigan
  - Haematology-Oncology Associates of Ohio and Michigan, PC, Lambertville, Michigan
  - Sparrow Regional Cancer Center, Lansing, Michigan
  - St. Mary Mercy Hospital, Livonia, Michigan
  - Community Cancer Center of Monroe, Monroe, Michigan
  - Mercy Memorial Hospital - Monroe, Monroe, Michigan
  - St. Joseph Mercy Oakland, Pontiac, Michigan
  - Mercy Regional Cancer Center at Mercy Hospital, Port Huron, Michigan
  - Seton Cancer Institute at Saint Mary's - Saginaw, Saginaw, Michigan
  - St. John Macomb Hospital, Warren, Michigan
  - MeritCare Bemidji, Bemidji, Minnesota
  - Duluth Clinic Cancer Center - Duluth, Duluth, Minnesota
  - CCOP - Duluth, Duluth, Minnesota
  - Miller - Dwan Medical Center, Duluth, Minnesota
  - Immanuel St. Joseph's, Mankato, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CCOP - MeritCare Hospital, Fargo, North Dakota
  - MeritCare Broadway, Fargo, North Dakota
  - Wood County Oncology Center, Bowling Green, Ohio
  - Hematology Oncology Center, Elyria, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - Northwest Ohio Oncology Center, Maumee, Ohio
  - St. Luke's Hospital, Maumee, Ohio
  - St. Charles Mercy Hospital, Oregon, Ohio
  - Toledo Clinic - Oregon, Oregon, Ohio
  - Firelands Regional Medical Center, Sandusky, Ohio
  - North Coast Cancer Care, Incorporated, Sandusky, Ohio
  - Flower Hospital Cancer Center, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - Toledo Hospital, Toledo, Ohio
  - St. Vincent Mercy Medical Center, Toledo, Ohio
  - Medical University of Ohio Cancer Center, Toledo, Ohio
  - CCOP - Toledo Community Hospital, Toledo, Ohio
  - Toledo Clinic, Incorporated - Main Clinic, Toledo, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - Fredericksburg Oncology, Incorporated, Fredericksburg, Virginia
  - Franciscan Skemp Healthcare - La Crosse Campus, La Crosse, Wisconsin

REFERENCES:
- [Background] Atherton PJ, Burger KN, Loprinzi CL, Neben Wittich MA, Miller RC, Jatoi A, Sloan JA. Using the Skindex-16 and Common Terminology Criteria for Adverse Events to assess rash symptoms: results of a pooled-analysis (N0993). Support Care Cancer. 2012 Aug;20(8):1729-35. doi: 10.1007/s00520-011-1266-x. Epub 2011 Sep 16. PMID 21922203
- [Result] Jatoi A, Dakhil SR, Sloan JA, Kugler JW, Rowland KM Jr, Schaefer PL, Novotny PJ, Wender DB, Gross HM, Loprinzi CL; North Central Cancer Treatment Group. Prophylactic tetracycline does not diminish the severity of epidermal growth factor receptor (EGFR) inhibitor-induced rash: results from the North Central Cancer Treatment Group (Supplementary N03CB). Support Care Cancer. 2011 Oct;19(10):1601-7. doi: 10.1007/s00520-010-0988-5. Epub 2010 Sep 6. PMID 20820817
- [Result] Jatoi A, Rowland K, Sloan JA, Gross HM, Fishkin PA, Kahanic SP, Novotny PJ, Schaefer PL, Johnson DB, Tschetter LK, Loprinzi CL. Tetracycline to prevent epidermal growth factor receptor inhibitor-induced skin rashes: results of a placebo-controlled trial from the North Central Cancer Treatment Group (N03CB). Cancer. 2008 Aug 15;113(4):847-53. doi: 10.1002/cncr.23621. PMID 18543329
- [Result] Jatoi A, Rowland K, Sloan JA, et al.: Does tetracycline prevent/palliate epidermal growth factor receptor (EGFR) inhibitor-induced rash? A phase III trial from the North Central Cancer Treatment Group (N03CB). [Abstract] J Clin Oncol 25 (Suppl 18): A-LBA9006, 494s, 2007.